CLINICAL TRIAL: NCT04084509
Title: Molecular and Functional Imaging of Parkinson's Pathology in SNCA, Parkin and PINK1 Mutation Carriers
Brief Title: Molecular and Functional Imaging in SNCA, Parkin and PINK1
Status: Withdrawn | Type: Observational
Why Stopped: Change of circumstances for CI/PI.
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: 263369
Record Dates: First submitted 2019-08-08; First posted 2019-09-10 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; PARK1; PARK2
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Controls
- Idiopathic Parkinson's Disease
- Symptomatic Genetic Carriers (SNCA, Parkin or PINK1)
- Asymptomatic Genetic Carriers (SNCA, Parkin or PINK1)

SUMMARY:
Parkinson's Disease (PD) is a progressive neurodegenerative disease characterized clinically by bradykinesia, resting tremor, rigidity, and postural instability. The hallmark pathophysiological alteration is a loss of dopaminergic transmission across the nigrostriatal pathway. According to Braak's neuropathological staging of disease, the pathological process in PD occurs in a gradual ascending fashion, starting from the olfactory bulb and progressing to the brainstem, with preferential involvement of the raphe nuclei, which contain serotonergic nuclei, and the noradrenergic locus coeruleus, before involving the substantia nigra and thereafter the whole brain. Little is known about the mechanisms underlying neuronal degeneration in PD and currently, no treatment is available to halt disease progression in PD. The pathophysiological characterisation of phenomena occurring in the time window between the pathological start of the disease and the onset of motor symptoms is crucial to develop potential neuroprotective agents. Several genes causing, the so-called monogenic parkinsonism, have been discovered providing important insights on the pathogenesis of PD.

The objective of the study is to characterize the molecular phenomena underlying genetic forms of parkinsonism and, therefore, providing further insights about the possible mechanisms taking place in PD and help identify targets for disease-modifying therapeutics, by using PET imaging with [11C]DASB (a marker of Serotonin transporter), SPECT imaging using [123I]FP-CIT (a marker of the presynaptic Dopamine transporter), and multi-modal MRI imaging, clinical markers (motor and non-motor symptoms and neuropsychological battery), blood and CSF biomarkers.

ELIGIBILITY:
Inclusion Criteria (for all subjects):

* All subjects must be judged by the investigator able to understand the nature, design, and procedures of the study and must be able to provide a signed and dated informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* All subjects must be willing and able to comply with scheduled visits, required study procedures and laboratory tests.
* All subjects must be able to travel to the research sites for the study procedures.
* For female subjects: They must be either of non-childbearing potential (either surgically sterile or post- menopausal - defined as 12 months of spontaneous amenorrhea), or, if of childbearing potential, subjects must demonstrate to be non-pregnant (as demonstrated by negative urine β-HCG test at screening), non-breastfeeding.
* All subjects must comply with highly effective contraceptive measures. A highly effective contraceptive measure is defined as a measure that can achieve a failure rate of less than 1% per year when used consistently and correctly. These methods are listed in more detail below:

Oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation;

Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation:

Intrauterine device (IUD) Intrauterine hormone-releasing system (IUS) Bilateral tubal occlusion Vasectomised partner Sexual abstinence

* For sexually active male subjects, they must agree to use condoms to protect their partners from becoming pregnant for the duration of the study and for 3 months after the last administration of PET or SPECT ligands. They must also agree to ensure that they and their partners are routinely using a medically approved contraceptive method. It is important that male subjects not impregnate others for the duration of the study and for 3 months after the last administration of PET or SPECT ligands.
* All subjects must have adequate visual and auditory acuity according to investigator's judgement to complete the psychological testing.
* All subjects must have no use of medications with known interaction with serotonergic transmission (e.g. selective serotonin reuptake inhibitors, tricyclic antidepressant, triptans, etc).
* For subjects taking any drugs that might interfere with dopamine transporter SPECT imaging (neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative) must be willing and able from a medical standpoint to hold the medication for at least 5 half-lives prior to screening DaTSCAN imaging.

Exclusion Criteria (for all subjects):

* Subjects lacking capacity according to investigator judgement.
* Subjects with a clinical diagnosis of dementia as determined by the investigator.
* Current treatment with anticoagulants (e.g. coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Use of any of the following drugs that might interfere with dopamine transporter SPECT imaging: neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 5 months of Screening.
* Use of investigational drugs or devices within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
* History of cancer within the last 5 years, with the exception of non-metastatic basal cell carcinoma of the skin.
* Subjects with current or recent history of drug or alcohol abuse/dependence.
* Contraindication to MRI, such as presence of metal devises or implants (e.g. pacemaker, vascular- or heart- valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes;
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable.
* Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls Idiopathic Parkinson's Disease Symptomatic Genetic Carriers (SNCA, Parkin or PINK1) Asymptomatic Genetic Carriers (SNCA, Parkin or PINK1)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes | Up to 21 days
  To quantify serotonergic and dopaminergic pathology in carriers of genetic mutations for familial forms of Parkinsonism, idiopathic PD patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politis, MD MSc PhD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided